CLINICAL TRIAL: NCT00539019
Title: Quantification and Derivation of Metabolic Needs in Children During Burn Rehabilitation
Status: Withdrawn | Type: Observational
Why Stopped: indirect calorimetry no longer employed at the institution; calorimeter is not accurate/reliable
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Theresa Mayes, Clinical Dietitian, Shriners Hospitals for Children
Other Study IDs: 05-11-17-03-EE
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Burns
Keywords: nutrition assessment; pediatric
MeSH Terms: conditions — Burns

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- A, observed: measure REE via indirect calorimetry at various time points post burn
  Interventions: Other: calories measured 5x following wound healing

INTERVENTIONS:
Other: calories measured 5x following wound healing — measure REE at various time points postburn

SUMMARY:
The investigators are collecting information on the calorie needs of patients in the first year postburn. The investigators hypothesize that increased energy needs continue for up to a year following wound closure from burn injury.

ELIGIBILITY:
Inclusion Criteria:

* >25% burn surface area
* Wounds present as 95% healed
* Admitted to Shriners Hospital Cincinnati within 7 days of injury

Exclusion Criteria:

* <5years old
* <25% burn injury
* admitted greater than 7 days postburn

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: burned, pediatrics pooled from inpatient acute population
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Theresa M Mayes, RD,LD, Principal Investigator — Shriners Hospital for Children, Cincinnati, Ohio
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States